CLINICAL TRIAL: NCT05677620
Title: Predictive Morphological Factors for Prescribing a Mandibular Advancement Device in the Therapeutic Approach of Obstructive Sleep Apnea
Brief Title: Predictive Factors for Prescribing a Mandibular Advancement Device for the Treatment of Obstructive Sleep Apnea
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Egas Moniz - Cooperativa de Ensino Superior, CRL (Other)
Collaborators: CUF Tejo Hospital (Unknown); Orthoapnea (Unknown)
Responsible Party: Sponsor
Other Study IDs: PHDPMC
Record Dates: First submitted 2022-12-15; First posted 2023-01-10 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Oral Appliance; DISE; Computed Tomography; Mandibular Advancement Device
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Propofol; Occlusal Splints

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Group A - Pharyngeal Computed Tomography Group: 22 randomly selected patients with mild to moderate obstructive sleep apnea will undergo pharyngeal CT with cephalometry and with registration in maximum comfortable protrusion (MCP)
  Interventions: Radiation: Pharyngeal Computed Tomography; Device: Mandibular Advancement Device
- Group B - Drug-Induced Sleep Endoscopy Group: 22 randomly selected patients with mild to moderate obstructive sleep apnea will undergo Drug-induced sleep endoscopy with registration in maximum comfortable protrusion (MCP)
  Interventions: Drug: Drug-Induced Sleep Endoscopy (Propofol); Device: Mandibular Advancement Device
- Group C - Pharyngeal Computed Tomography and Drug-Induced Sleep Endoscopy Group: 22 randomly selected patients with mild to moderate obstructive sleep apnea will undergo a pharyngeal computed tomography + Drug-induced sleep endoscopy with registration in maximum comfortable protrusion (MCP)
  Interventions: Radiation: Pharyngeal Computed Tomography; Drug: Drug-Induced Sleep Endoscopy (Propofol); Device: Mandibular Advancement Device

INTERVENTIONS:
Radiation: Pharyngeal Computed Tomography — To assess the presence of a possible level/level of collapse, a pharyngeal CT with cephalometry will be performed, and a standard classification system, VOTE, will be used. After obtaining said CT, the dentist will place the recording in MCP and perform a new CT scan of the pharynx with cephalometry and with the MCP recording set intraorally to assess whether this position reduces or eliminates the collapse from UA.
  Other Names: Pharyngeal CT
  Groups: Group A - Pharyngeal Computed Tomography Group; Group C - Pharyngeal Computed Tomography and Drug-Induced Sleep Endoscopy Group
Drug: Drug-Induced Sleep Endoscopy (Propofol) — The DISE technique will be performed by an otorhinolaryngologist (ENT) with a nasopharyngoscope in a operating room. This technique is complemented with bite registration (MCP). Artificial sleep will be induced by intravenous administration of propofol through an infusion system controlled by an anesthesiologist (2.0-3.0 mcg/mL). The following variables will be continuously monitored: electrocardiography, oxygen saturation, and bispectral index (BIS). In this phase of the DISE, the upper airways will be evaluated during sleep with the MCP positioned intra-orally.
  Other Names: DISE
  Groups: Group B - Drug-Induced Sleep Endoscopy Group; Group C - Pharyngeal Computed Tomography and Drug-Induced Sleep Endoscopy Group
Device: Mandibular Advancement Device — A duo-block, titratable, and customized MAD (NOA®; Orthoapnea) will be fitted for each patient who starts treatment with MAD. The MAD consists of two CAD/CAM polyamide intraoral devices (one for the upper and one for the lower arch). The adaptation period takes place over one month. After this adaptation, patients will undergo a new PSG using MAD.
  Other Names: MAD

SUMMARY:
This project evaluates the morphological predictive factors for prescribing a mandibular advancement device in the therapeutic approach of Obstructive sleep apnea (OSA). The investigators will carry out the project with patients who travel to CUF Tejo Hospital to solve their sleep disturbance, namely cases of obstructive sleep apnea. The investigators designed three groups of 22 individuals each. The investigators will only include individuals after signing the informed consent. In the 1st appointment, the principal investigator will conduct a complete anamnesis and a clinical examination, where several items will be documented: Age, gender, body mass index, mallampati index, neck, and waist circumference. The clinical interview will assess the patient's daytime sleepiness, nighttime snoring, and quality of life through the respective questionnaires: the Epworth Sleepiness Scale (ESS), the snoring severity scale (SSS), and the Sleep Apnea Quality of Life Index (SAQLI). Still, in the 1st consultation, a level III Polysomnography (PSG) will be prescribed to assess the possibility of OSA, and a pharyngeal computed tomography (CT) with cephalometric analysis and recording in maximum comfortable protrusion to evaluate the Upper Airway (UA) and the prognosis of mandibular advancement in case of UA collapse. The other group will perform Drug-Induced Sleep Endoscopy (DISE) and CT with registration in maximum comfortable protrusion. Then, the investigators will make personalized and titled mandibular advancement devices (MAD). The measurements and PSG III questionnaires will be carried out after 1 and 6 months to evaluate the results.

DETAILED DESCRIPTION:
This study will present 66 adult patients diagnosed with mild or moderate OSA (5 <AHI ≤ 30/h) through polysomnography (PSG) level III, referred from pulmonology, otorhinolaryngology and/or neurology for treatment with MAD, who refuse or do not tolerate the therapeutic approach of CPAP, in the sleep unit of Hospital CUF Tejo. The randomization sequence will be generated by computer and kept confidential, in a sealed and opaque envelope, until the moment of recruitment. There will be 3 study groups:

Group A - Will perform pharyngeal CT with cephalometry and registration in maximum comfortable protrusion (MCP).

Group B - Will perform the DISE with registration in MCP. Group C - Will perform pharyngeal CT with cephalometry and recording in MCP + DISE with recording in MCP

In the first appointment, a complete anamnesis and a clinical examination will be carried out, where several items will be documented: Age, gender, BMI, mallampati index, neck, and waist circumference. The clinical interview will assess daytime sleepiness, nighttime snoring, and the patient's quality of life through the respective questionnaires: the Epworth Sleepiness Scale (ESS), the snoring severity scale (SSS), and the Sleep Apnea Quality of Life Index (SAQLI). Using a Likert scale, the ESS is a quantitative assessment tool for drowsiness or the propensity to fall asleep in eight everyday situations. This instrument has been used in various contexts, populations, and clinical conditions, emphasizing sleep-disordered breathing, namely OSA. The SSS is a three-question questionnaire that assesses the intensity, frequency, and duration of snoring, completed by patients and their bed partners. The SSS is internally consistent across patients, regardless of age and sex, and externally valid, as it has a high correlation with the respiratory disturbance index (RDI), AHI, and ESS. The SAQLI was created as a specific quality-of-life instrument for patients with OSAS. This is a 35-item questionnaire that assesses the adverse impact of OSA in four domains: daily animosity, social interactions, emotional state, and symptoms. Items are scored on a 7-point scale. Still, in the 1st consultation, a PSG level III will be prescribed to assess the possibility of OSA and a CT of the pharynx with cephalometric analysis and recording in MCP to assess the UA and the prognosis of advancement of the mandible in the UA collapse/s.

After confirmation of mild to moderate OSA and application of the inclusion and exclusion criteria, patients will be randomly allocated into 3 study groups, with the randomization sequence generated by computer and kept secret in a sealed and opaque envelope until the time of recruitment:

Group A - Will undergo CT of the pharynx with cephalometry and recording in MCP and will be evaluated as a "poor candidate," "candidate with a moderate resolution," or "good candidate." Group B - Will perform the DISE with registration in MCP and will be evaluated as a "bad candidate," "candidate with a moderate resolution," or "good candidate." Group C - Will undergo pharyngeal CT with cephalometry and recording in MCP + DISE with MCP recording and will be evaluated as a "bad candidate," "candidate with a moderate resolution," or "good candidate."

In the second appointment, impressions will be made for the MAD, and in the third appointment, the MAD will be delivered.

After one month of use and adaptation to the MAD, the three groups will perform a PSG level III, in which the patient will have the MAD placed intra-orally, and the ESS, SSS, and SAQLI questionnaires will be filled out again, and the evaluation of adaptation to the MAD will be carried out (self-report).

After six months of using the MAD, the three groups will again perform a PSG level III, in which the patient will have the DAM placed intra-orally in the same mandibular advancement position that was placed in the previous follow-up. The ESS questionnaires will be completed, including SSS, SAQLI, and assessment of adaptation to the MAD (self-report).

The objective treatment outcome will be based on the PSG level III results with the MAD. An effective response to treatment will be defined as a reduction in AHI after treatment with MAD of 50% compared to baseline, and non-response will be described as a reduction in AHI of <50%. For patients who do not present an effective response in the 1st Follow-up (where PSG level III will be performed one month after adaptation to the MAD), the MAD will be titrated (with more significant mandibular advancement) with the aim of, in the 2nd Follow-up up (where PSG level III will be performed six months after adaptation to the MAD) to obtain an adequate response, always thinking about the most significant possible AHI reduction to improve the patient's quality of life. It will also be analyzed whether the assessment during DISE, that the patient is a "good candidate," "candidate with a moderate resolution," and "poor candidate," is effective after PSG with MAD.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 70 years of age with the indication for treatment with mandibular advancement device, who refused or cannot tolerate CPAP;
* Body Mass Index (BMI) between 19 and 34.9 Kg/m2;
* The presence of 8 healthy teeth or more per jaw (upper and lower );
* Maximum mandibular protrusion capacity of at least 6 mm.

Exclusion Criteria:

* Significant nasal obstruction; chronic lung disease;
* Class III or IV congestive heart failure according to the New York Heart Association classification;
* Neuromuscular diseases or previous upper airway surgery unrelated to obstructive sleep apnea;
* Uncontrolled periodontitis;
* Tooth mobility;
* Orthodontic treatment;
* Dental prosthesis wholly or partially removable.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will present 66 adult patients diagnosed with mild or moderate OSAS (5 <AHI ≤ 30/h) through polysomnography (PSG) level III, referred from pulmonology, otorhinolaryngology and/or neurology for treatment with ADM, who refuse or do not tolerate the therapeutic approach of CPAP, in the sleep unit of Hospital CUF Tejo.
Sampling Method: Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Changes in the apnea-hypopnea index | Before making and starting to use the MAD and one and six months after
  The apnea-hypopnea index will be registered with the level III polysomnography and we will evaluate after using the MAD if there were improvements or not, relating to the predictors that we analyzed before.
Changes in upper airway collapse analyzed by CT Pharyngeal | Through study completion, an average of six months
  the prognosis for the use of a MAD using the MCP recording and VOTE scoring system: when the upper airway collapse has entirely resolved (no residual collapse at any level of the upper airway), with the bite registration in MCP, the patient will be considered a "Good Candidate." Suppose there is only partial resolution (improvement, but with the residual or multilevel collapse of the upper airway) with the bite registration in PMC. In that case, you will qualify as a "moderately resolved candidate." If upper airway collapse remains unchanged or worsens with PMC bite registration, patients will be considered a "poor candidate."
Changes in Upper Airway collapse analyzed by DISE | through study completion, an average of six months
  Evaluation of the prognosis for the use of a MAD, we will use the mandibular advancement record in MCP. The VOTE classification: when the UA collapse is completely resolved (no residual collapse at any level of the upper airway), and there is no snoring, with the bite registration in MCP, the patient will be considered a "Good Candidate." Suppose there is only partial resolution (improvement, but with the residual or multilevel collapse of the UA) and some snoring with the bite registration in MCP. In that case, he will qualify as a "candidate with moderate resolution." If UA collapse remains unchanged or worsens with MCP bite registration and still snoring, patients will be considered a "bad candidate."

SECONDARY OUTCOMES:
Subjective assessment of daytime sleepiness | Before making and starting to use the MAD and one and six months after
  The subjective evaluation will be done through a validated questionnaire: Epworth Sleepiness Scale (ESS). The ESS asks the respondent to rate on a 4-point scale (0-3). The higher the score, the more severe the daytime sleepiness
Subjective assessment of quality of life | Before making and starting to use the MAD and one and six months after
  The subjective evaluation will be carried out through a validated questionnaire - Sleep Apnea Quality of Life Index (SAQLI) -a 35-item questionnaire that assesses the adverse impact of OSA. Items are scored on a 7-point scale.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Manso, PhD, Study Director — Egas Moniz School of Health and Science
Locations (1):
- CUF Tejo Hospital, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.